CLINICAL TRIAL: NCT06150118
Title: The Effect of Cognitive Behavioral Therapy and Virtual Reality Use in Supporting Physical Rehabilitation After Anterior Cruciate Ligament (ACL) Operation: A Parallel-Arm Randomized Controlled Trial
Brief Title: The Effect of Cognitive Behavioral Therapy and Virtual Reality Use in Inured Athletes
Acronym: CBT+VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Hande Turkeri Bozkurt, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 121K248
Record Dates: First submitted 2023-11-17; First posted 2023-11-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Re-injury Anxiety; Kinesiophobia; Poor Rehabilitation Adherence; Poor Rehabilitation Self Efficacy; Return to Sport
Keywords: Re-injury anxiety; Adherence; Self-efficacy; Kinesiophobia; psychological readiness to return to sport
MeSH Terms: conditions — Kinesiophobia | interventions — Cognitive Behavioral Therapy; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CBT+VR (Cognitive behavioral therapy and virtual reality) (Experimental)
  Interventions: Other: CBT+VR (Cognitive behavioral therapy and virtual reality)
- Control (Placebo Comparator)
  Interventions: Behavioral: Control (placebo) group
- Control Group (No Intervention): This arm have no intervention during the research. They only had been followed up by researchers
- CBT (Cognitive Behavioral Therapy) (Experimental)
  Interventions: Other: CBT (Cognitive Behavioral Therapy)
- VR (Virtual reality) (Experimental)
  Interventions: Behavioral: VR (Virtual reality)

INTERVENTIONS:
Other: CBT+VR (Cognitive behavioral therapy and virtual reality) — The investigators are testing whether this intervention protocol is effective on re-injury anxiety, kinesiophobia, self-efficacy, and adherence problems in athletes who have undergone ACL surgery.
  Arms: CBT+VR (Cognitive behavioral therapy and virtual reality)
Behavioral: Control (placebo) group — The investigators are testing whether the placebo control protocol is effective on re-injury anxiety, kinesiophobia, self-efficacy, and adherence problems in athletes who have undergone ACL surgery.
  Arms: Control
Behavioral: VR (Virtual reality) — The investigators are testing whether this intervention protocol is effective on re-injury anxiety, kinesiophobia, self-efficacy, and adherence problems in athletes who have undergone ACL surgery.
  Arms: VR (Virtual reality)
Other: CBT (Cognitive Behavioral Therapy) — The investigators are testing whether this intervention protocol is effective on re-injury anxiety, kinesiophobia, self-efficacy, and adherence problems in athletes who have undergone ACL surgery.
  Arms: CBT (Cognitive Behavioral Therapy)

SUMMARY:
In this study, which aimed to develop a Cognitive Behavioral Therapy (CBT) protocol enriched with Virtual Reality (VR) to address the psychological responses that arise after ACL surgery, and to examine the effectiveness of this protocol. The effectiveness of the protocol was assessed using pre-test, post-test, and two follow-up measurements with the Re-Injury Anxiety Inventory (RIAI), the Sport Injury Rehabilitation Adherence Scale (SIRAS), the Tampa Scale for Kinesiophobia (TSK), the Athletic Injury Self-Efficacy Questionnaire (AISEQ), the Return to Sport After Serious Injury Questionnaire (RSSIQ), and the Anterior Cruciate Ligament Return to Sport Scale (ACL-RSI). Anxiety levels during VR exposure sessions were measured through biofeedback and the Subjective Units of Distress Scale (SUDS).

DETAILED DESCRIPTION:
In this study, which aimed to develop a Cognitive Behavioral Therapy (CBT) protocol enriched with Virtual Reality (VR) to address the psychological responses that arise after ACL surgery, and to examine the effectiveness of this protocol. The protocol was developed in 5 stages and a randomized controlled trial was conducted with 60 athletes to test its effectiveness. The study consisted of 3 experimental and 2 control groups. One of the control group was a plasebo control group.The effectiveness of the protocol was assessed using pre-test, post-test, and follow-up measurements with the Re-Injury Anxiety Inventory (RIAI), the Sport Injury Rehabilitation Adherence Scale (SIRAS), the Tampa Scale for Kinesiophobia (TSK), the Athletic Injury Self-Efficacy Questionnaire (AISEQ), the Return to Sport After Serious Injury Questionnaire (RSSIQ), and the Anterior Cruciate Ligament Return to Sport Scale (ACL-RSI). Anxiety levels during VR exposure sessions were measured through biofeedback and the Subjective Units of Distress Scale (SUDS).

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Have had an ACL injury operation
* Be between the ages of 18 and 45
* To be a professional athlete in Turkish leagues
* Being an athlete in football, volleyball, and basketball

Exclusion Criteria:

* Having a discomfort that prevents participants from participating in VR sessions (panic attack, epilepsy, etc.)
* Having decided to quit sports even if participants will continue rehabilitation after the operation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Re-Injury Anxiety Inventory (RIAI) | Through study completion, an average of 1 year
  This scale measures re-injury anxiety
Sport Injury Rehabilitation Adherence Scale (SIRAS) | Through study completion, an average of 1 year
  This scale measures rehabilitation adherence
Athletic Injury Self-Efficacy Questionnaire (AISEQ) | Through study completion, an average of 1 year
  This scale measures Self-Efficacy
Tampa Scale for Kinesiophobia | Through study completion, an average of 1 year
  This scale measures kinesiophobia
Return to Sport After Serious Injury Questionnaire (RSSIQ) | Through study completion, an average of 1 year
  This scale was used to assess whether athletes were psychologically ready to return to sport.
Anterior Cruciate Ligament Return to Sport Scale (ACL-RSI) | Through study completion, an average of 1 year
  This scale was used to assess whether athletes were psychologically ready to return to sport from ACL surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ziya Koruç, PhD, Study Director — Hacettepe University; Britton W. Brewer, PhD, Study Director — Springfield College
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No